CLINICAL TRIAL: NCT05761574
Title: A Full-Factorial, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Single-Dose Efficacy and Safety Study of an Acetaminophen/Naproxen Sodium Fixed Combination, Acetaminophen, and Naproxen Sodium in Postoperative Dental Pain
Brief Title: A Study of an Acetaminophen/Naproxen Sodium Fixed Combination, Acetaminophen and Naproxen Sodium in Postoperative Dental Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CCSPAA005199; CCSPAA005199 (Other Grant/Funding Number: Johnson & Johnson Consumer, Inc. (JJCI))
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-05

CONDITIONS: Pain
Keywords: Analgesics; Dental Pain; Acetaminophen; Naproxen Sodium; Pain; Fixed-Dose
MeSH Terms: conditions — Pain; Toothache | interventions — Acetaminophen; Naproxen

STUDY DESIGN:
Intervention Model Description: Post-operative dental pain following third molar extraction.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Acetaminophen/Naproxen Sodium Fixed Combination (Experimental): Participants will receive a single oral dose of two Acetaminophen/Naproxen Sodium Fixed Combination tablets.
  Interventions: Drug: Acetaminophen/Naproxen Sodium Fixed Combination
- Naproxen Sodium (Active Comparator): Participants will receive a single oral dose of one Naproxen Sodium tablet with one Placebo capsule.
  Interventions: Drug: Naproxen Sodium; Drug: Placebo
- Acetaminophen (Active Comparator): Participants will receive a single oral dose of two Acetaminophen tablets.
  Interventions: Drug: Acetaminophen
- Placebo (Placebo Comparator): Participants will receive a single oral dose of two Placebo capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetaminophen/Naproxen Sodium Fixed Combination — Fixed combination of Acetaminophen/Naproxen Sodium will be administered orally.
  Arms: Acetaminophen/Naproxen Sodium Fixed Combination
Drug: Naproxen Sodium — Naproxen Sodium will be administered orally.
  Arms: Naproxen Sodium
Drug: Acetaminophen — Acetaminophen will be administered orally.
  Arms: Acetaminophen
Drug: Placebo — Placebo will be administered orally.
  Arms: Naproxen Sodium; Placebo

SUMMARY:
The purpose of this study is to evaluate how well a fixed combination of acetaminophen/naproxen sodium relieves postoperative dental pain compared with acetaminophen, naproxen sodium and placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single-dose full-factorial study to evaluate the analgesic efficacy and safety of a fixed combination of acetaminophen and naproxen sodium, compared with acetaminophen or naproxen sodium alone, and placebo following surgical extraction of three or four third molars.

ELIGIBILITY:
Inclusion Criteria:

* Weigh 100 pounds or greater and have a body mass index (BMI) of 17.5 to 30.4 (inclusive) at screening
* Surgical removal of three or four third molars, of which, two must be mandibular impactions
* Meets requirements for post-surgical pain level
* Females of childbearing potential and males agree to contraceptive requirements of study
* Have a negative urine drug screen at screening, and on day of surgical procedure

Exclusion Criteria:

* Pregnant female, breastfeeding, trying to become pregnant or male with pregnant partner or partner currently trying to become pregnant
* Have a known allergy or hypersensitivity to naproxen (or other NSAIDs including aspirin) or to acetaminophen, oxycodone or other opioids
* Not able to swallow whole large tablets or capsules
* History of any condition(s) in investigator's opinion, may jeopardize subject safety, well-being and integrity of study
* Use analgesics 5 or more times per week
* History of chronic tranquilizer use, heavy drinking, or substance abuse, as judged by the investigator site staff, in the last 5 years
* Use any immunosuppressive drugs within 2 weeks of surgical procedure
* History of endoscopically documented peptic ulcer disease or bleeding disorder in the last 2 years

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 447 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Time-weighted Sum of Pain Intensity Difference from 0 to 12 Hours After Dosing (SPID 0-12) | 0 to 12 hours
  Time-weighted sum of pain intensity difference (SPID) scores will be calculated using values collected on the Pain Intensity-Numerical Rating Scale (PI-NRS) ranging from 0-10 (0 = no pain, 10 = very severe pain) collected at each scheduled timepoint within the specified timeframe.

SECONDARY OUTCOMES:
Time-weighted Sum of Pain Intensity Difference From 6 to 12 Hours (SPID 6-12) | 6 to 12 hours
  Time-weighted sum of pain intensity difference (SPID) scores will be calculated using values collected on the PI-NRS ranging from 0-10 (0 = no pain, 10 = very severe pain) collected at each scheduled timepoint within the specified timeframe.
Time to First Request of Rescue Analgesic | 0 to 24 hours
  Time to first request for rescue medication will be measured as the elapsed time from when investigational product (IP) was given until the time rescue medication was first requested.
Percentage of Participants who Request Rescue Analgesic During the First 12 hours | 0 to 12 hours
  Percentage of participants who request rescue analgesic during the first 12 hours will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bertoch, Principal Investigator — JBR Clinical Research
Locations (1):
- JBR Clinical Research LLC, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] GUZMAN F, BRAUN C, LIM RK, POTTER GD, RODGERS DW. NARCOTIC AND NON-NARCOTIC ANALGESICS WHICH BLOCK VISCERAL PAIN EVOKED BY INTRA-ARTERIAL INJECTION OF BRADYKININ AND OTHER ALGESIC AGENTS. Arch Int Pharmacodyn Ther. 1964 Jun 1;149:571-88. No abstract available. PMID 14191090
- [Background] LIM RK, GUZMAN F, RODGERS DW, GOTO K, BRAUN C, DICKERSON GD, ENGLE RJ. SITE OF ACTION OF NARCOTIC AND NON-NARCOTIC ANALGESICS DETERMINED BY BLOCKING BRADYKININ-EVOKED VISCERAL PAIN. Arch Int Pharmacodyn Ther. 1964 Nov 1;152:25-58. No abstract available. PMID 14248351
- [Background] Aronoff DM, Oates JA, Boutaud O. New insights into the mechanism of action of acetaminophen: Its clinical pharmacologic characteristics reflect its inhibition of the two prostaglandin H2 synthases. Clin Pharmacol Ther. 2006 Jan;79(1):9-19. doi: 10.1016/j.clpt.2005.09.009. No abstract available. PMID 16413237
- [Background] Pickering G, Loriot MA, Libert F, Eschalier A, Beaune P, Dubray C. Analgesic effect of acetaminophen in humans: first evidence of a central serotonergic mechanism. Clin Pharmacol Ther. 2006 Apr;79(4):371-8. doi: 10.1016/j.clpt.2005.12.307. PMID 16580905
- [Background] Mallet C, Daulhac L, Bonnefont J, Ledent C, Etienne M, Chapuy E, Libert F, Eschalier A. Endocannabinoid and serotonergic systems are needed for acetaminophen-induced analgesia. Pain. 2008 Sep 30;139(1):190-200. doi: 10.1016/j.pain.2008.03.030. Epub 2008 May 15. PMID 18485596
- [Background] Koch-Weser J. Drug therapy. Acetaminophen. N Engl J Med. 1976 Dec 2;295(23):1297-300. doi: 10.1056/NEJM197612022952306. No abstract available. PMID 790189
- [Background] Milton AS. Modern views on the pathogenesis of fever and the mode of action of antipyretic drugs. J Pharm Pharmacol. 1976 Apr;28(4 SUPPL):393-9. doi: 10.1111/j.2042-7158.1976.tb04186.x. No abstract available. PMID 6743
- [Background] Ameer B, Greenblatt DJ. Acetaminophen. Ann Intern Med. 1977 Aug;87(2):202-9. doi: 10.7326/0003-4819-87-2-202. PMID 329728
- [Background] Product Monograph for Aleve (Naproxen Sodium Tablets USP/Liquid Gels/Capsules 220 mg). Bayer Inc. Consumer Care. Revised 8 January 2015
- [Background] Todd PA, Clissold SP. Naproxen. A reappraisal of its pharmacology, and therapeutic use in rheumatic diseases and pain states. Drugs. 1990 Jul;40(1):91-137. doi: 10.2165/00003495-199040010-00006. PMID 2202585
- [Background] Davies NM, Anderson KE. Clinical pharmacokinetics of naproxen. Clin Pharmacokinet. 1997 Apr;32(4):268-93. doi: 10.2165/00003088-199732040-00002. PMID 9113437
- [Background] Cooper SA, Desjardins PJ. The value of the dental impaction pain model in drug development. Methods Mol Biol. 2010;617:175-90. doi: 10.1007/978-1-60327-323-7_15. PMID 20336423
- [Background] Cooper SA, Desjardins PJ, Turk DC, Dworkin RH, Katz NP, Kehlet H, Ballantyne JC, Burke LB, Carragee E, Cowan P, Croll S, Dionne RA, Farrar JT, Gilron I, Gordon DB, Iyengar S, Jay GW, Kalso EA, Kerns RD, McDermott MP, Raja SN, Rappaport BA, Rauschkolb C, Royal MA, Segerdahl M, Stauffer JW, Todd KH, Vanhove GF, Wallace MS, West C, White RE, Wu C. Research design considerations for single-dose analgesic clinical trials in acute pain: IMMPACT recommendations. Pain. 2016 Feb;157(2):288-301. doi: 10.1097/j.pain.0000000000000375. PMID 26683233
- [Background] Lipkovich I, Ratitch B, O'Kelly M. Sensitivity to censored-at-random assumption in the analysis of time-to-event endpoints. Pharm Stat. 2016 May;15(3):216-29. doi: 10.1002/pst.1738. Epub 2016 Mar 21. PMID 26997353
- [Background] Cheung R, Krishnaswami S, Kowalski K. Analgesic efficacy of celecoxib in postoperative oral surgery pain: a single-dose, two-center, randomized, double-blind, active- and placebo-controlled study. Clin Ther. 2007;29 Suppl:2498-510. doi: 10.1016/j.clinthera.2007.12.008. PMID 18164917
- [Background] Fricke J, Davis N, Yu V, Krammer G. Lumiracoxib 400 mg compared with celecoxib 400 mg and placebo for treating pain following dental surgery: a randomized, controlled trial. J Pain. 2008 Jan;9(1):20-7. doi: 10.1016/j.jpain.2007.08.004. Epub 2007 Oct 15. PMID 17933588
- [Background] Clinical Study Report CCSPAA001068. A randomized, double-blind, placebo- and activecontrolled, proof of concept study to evaluate two strengths of concomitantly dosed naproxen sodium with acetaminophen, compared with naproxen sodium, hydrocodone/acetaminophen and placebo in postoperative dental pain.: Johnson & Johnson Consumer, Inc., May 2019.
- [Background] Clinical Study Report CCSPAA002398. A Randomized, Double-blind, Placebo-controlled Study to Evaluate Five Strengths of a Fixed Combination of Acetaminophen/Naproxen Sodium in Postoperative Dental Pain.: Johnson & Johnson Consumer, Inc., November 2020.
- [Background] 21 CFR § 300.50 - Fixed-combination prescription drugs for humans, 40 FR 13496, Mar. 27, 1975, as amended at 64 FR 401, Jan. 5, 1999.
- [Background] Little RJ, Rubin DB. Statistical analysis with missing data: John Wiley & Sons; 2002.